CLINICAL TRIAL: NCT02928536
Title: The TackSHS Survey: a Cross-sectional Study on Secondhand Smoke in 12 European Countries
Brief Title: The TackSHS Survey: a Pan-European Study on SHS
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Institut Català d'Oncologia (Other); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: 6895
Record Dates: First submitted 2016-10-04; First posted 2016-10-10 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Second Hand Tobacco Smoke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — This is an observational study. No intervention is considered

SUMMARY:
Within the TackSHS project (H2020 project grant agreement No 681040), we will conduct a European cross-sectional study, aiming at i) estimating prevalence and investigating determinants of smoking, e-cigarette use and exposure to SHS and to e-cigarette aerosol; ii) analyzing the attitudes, perceptions and behaviours of the adult European population towards policies to limit SHS exposure; iii) comparing selected smoking-related data between TackSHS and a previously conducted pan-European survey; iv) assessing mortality and morbidity from selected respiratory and cardiovascular diseases attributable to SHS exposure among adults and children in Europe; v) quantifying the economic burden associated to the exposure to SHS and e-cigarette aerosol in Europe. Overall, approximately 12,000 individuals aged 15 years or over will be enrolled in 12 different European countries (BG, DE, ES, FR, GR, IE, IT, LV, PL, PT, RO, UK). Surveys will be representative of the country-specific population in terms of sex, age, and socio-economic characteristics.

DETAILED DESCRIPTION:
Study characteristics The TackSHS survey is a face-to-face population-based cross-sectional survey that will be conducted in 12 selected European countries, coordinated by Dr Silvano Gallus, Department of Epidemiology of the "Mario Negri" Institute (Milan, Italy).

Background Exposure to secondhand smoke (SHS) has serious adverse health effects on adults and children, causing more than 600,000 deaths each year worldwide. Estimates of prevalence of non-smokers exposed to SHS range between 20% and 60% in various European countries. The WHO recommend to develop smoke-free policies to protect non-smokers from SHS exposure. E-cigarettes have irrupted in the market over the last 5 years, and their sales and popularity have considerably grown in the European Union (EU). Approximately 7% of Europeans ever used e-cigarettes. TackSHS is a new research project funded by the European Commission (EC) within the Horizon 2020 programme (grant agreement: 681040). Within the TackSHS Project, selected work packages (WP; i.e., WP3, WP9 and WP10) involve the conduction of a survey in 12 EU countries: the TackSHS survey.

Objectives Objectives of this cross-sectional study include: i) to estimate prevalence, and investigate individual-level and country-specific determinants, of smoking, e-cigarette use, and exposure to SHS and to e-cigarette aerosol in selected European countries (WP3); ii) to analyze the attitudes, perceptions and behaviours of the adult European population towards policies to limit SHS exposure (WP3); iii) to compare selected smoking-related data collected through the TackSHS survey with those from a companion pan-European survey conducted in 2010 (WP3); iv) to assess morbidity and mortality from selected respiratory and cardiovascular diseases attributable to SHS exposure among adults and children in the European population (WP9); v) to quantify the economic burden associated to the exposure to SHS and e-cigarette aerosol in Europe (WP10).

Methods The cross-sectional survey will be conducted in 12 European countries (Bulgaria, England, France, Germany, Greece, Ireland, Italy, Latvia, Poland, Portugal, Romania, and Spain), representing geographical, legislative and cultural variations across the EU. In each of the 12 selected countries, approximately 1000 individuals, representative of the general population aged 15 years and over will be enrolled. The final sample will therefore include a total of approximately 12,000 subjects. The sample size in each specific country will allow us to obtain prevalence estimates with a maximum standard error (SE) lower than ± 1.6%. Therefore, with such a sample size we will be able to provide stable prevalence estimates (with a relatively small 95% confidence interval), overall, but also in each specific country.

Survey participants will have to satisfy the following inclusion criteria: i) 15 years and over of age; ii) residence in one of the 12 selected countries; iii) ability to understand and answer the questions of the questionnaire of the study in the country-specific language; iv) formal acceptance to participate in the study.

The multi-stage methodology will be used as the preferred sampling methodology, but other methods, including stratified or simple sampling or quota methods, will also be accepted wherever it is not possible to conduct a multistage random sampling.

Participants will be surveyed by trained interviewers through face-to-face interviews using a structured standardized questionnaire, including information on: i) socio-economic and demographic characteristics; ii) cigarette smoking habit and e-cigarette use; iii) SHS and e-cigarette aerosol exposures in different sites; iv) attitudes and perceptions on smoke-free regulations. Whenever possible, data will be collected within computer assisted personal interviews (CAPI). Alternatively, paper and pencil (P&P) interviews will be accepted.

Once the fieldwork is completed, data will be checked for coherence and for the presence of possible errors, cleaned, and finalized into a single dataset by expert biostatisticians at the Department of Epidemiology of "Mario Negri" Institute.

According to the statistical analyses, within WP3 both univariate and multivariate (i.e., multiple logistic regression) analyses will be considered to identify sub-groups of the population or clusters of countries more frequently exposed to SHS or to passive exposure to emissions from e-cigarettes. Moreover, to evaluate the changes in time of selected smoking-related aspects, TackSHS data will be compared with data from a previous companion European survey (the PPACTE survey). Within WP9, through the use of specific algorithms, it will be possible to estimate attributable mortality and morbidity to SHS in Europe, taking advantage of: i) prevalence figures on tobacco smoking and SHS exposure from the ThackSHS survey and other selected European datasets; ii) morbidity and mortality figures from the WHO and other sources; iii) and the quantification of the association between SHS exposure and the risk of SHS-related diseases from scientific literature reviews. Within WP10, using SHS exposure figures from the TackSHS survey, a Return On Investment model will be developed to assess the cost-effectiveness, budget impact and a wider set of social return on investment metrics of selected policies aimed at reducing exposure to SHS across European countries.

Ethical Issues Although in EU countries, according to their current legislation, it is not mandatory for this type of studies (i.e., population-based cross-sectional survey) to obtain either a formal approval of the study protocol from ethics committees or the written consent signed by survey participants, following the request of the European Commission, we will satisfy these both these ethical requirements. Thus, after evaluation of the Italian Ethics Committee (i.e., the Ethics Committee of the study coordinator), the study protocol will be submitted for evaluation to the Ethics Committees of the other 11 countries where data will be collected. Moreover, formal consent (and signature in case of P&P interview) will be obtained from each adult participant, and, in case of minors from one of their parents or legal tutors. All data will be managed anonymously, in respect of the privacy regulations in force, only for scientific purposes, without any lucrative aim. These and other measures are in agreement with national and current or forthcoming EU (i.e., Directive 95/46/EC) regulations.

Relevance, implications and dissemination Thanks to the TackSHS survey, we will provide a characterization of exposure to SHS and to e-cigarette aerosol in populations with different socioeconomic level and from various European countries. We will also provide the first estimates of morbidity and mortality due to SHS exposure at the European level, and the cost impact of interventions to control SHS exposure through purpose-built economic models. The main findings of the TackSHS survey will be disseminated on international peer-reviewed open-access journals and on the TackSHS Project website (www.tackshs.eu), and will be presented in national or international conferences.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 15 years and over;
* individuals resident of the 12 selected countries;
* individuals able to understand and answer the questions of the questionnaire of the study in the country-specific language;
* individuals who formally accept to participate in the study.

Exclusion Criteria:

No specific exclusion criteria are considered.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In each of the 12 selected European countries, approximately 1000 individuals, representative of the general population aged 15 years and over in terms of age, sex, geographic area, and socio-economic characteristics, will be enrolled in this cross-sectional study. The final sample will therefore include a total of approximately 12,000 subjects.
  Sample size computation The sample size in each specific country will allow us to obtain prevalence estimates with a maximum standard error (SE) lower than ± 1.6%. Therefore, with such a sample size we will be able to provide stable prevalence estimates (with a relatively small 95% confidence interval), overall but also in each specific country.
Sampling Method: Probability Sample
Enrollment: 11902 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvano Gallus, Sc.D, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- DOXA Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
No plan is made to share IPD. Main results (aggregated data) will be published in peer-reviewed open-access journals

REFERENCES:
- [Background] Fernandez E, Lopez MJ, Gallus S, Semple S, Clancy L, Behrakis P, Ruprecht A, Gorini G, Lopez-Nicolas A, Radu-Loghin C, Soriano JB; TackSHS Project Investigators; TackSHS Project Investigators. Tackling second-hand exposure to tobacco smoke and aerosols of electronic cigarettes: the TackSHS project protocol. Gac Sanit. 2020 Jan-Feb;34(1):77-82. doi: 10.1016/j.gaceta.2019.07.002. Epub 2019 Sep 23. PMID 31558386
- [Derived] Amalia B, Liu X, Lugo A, Fu M, Odone A, van den Brandt PA, Semple S, Clancy L, Soriano JB, Fernandez E, Gallus S; TackSHS Project Investigators. Exposure to secondhand aerosol of electronic cigarettes in indoor settings in 12 European countries: data from the TackSHS survey. Tob Control. 2021 Jan;30(1):49-56. doi: 10.1136/tobaccocontrol-2019-055376. Epub 2020 Mar 2. PMID 32123139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A pilot study was conducted in Italy in November 2016. The fieldwork in other countries was conducted between June 2017 (in Romania) and October 2018 (in Latvia). The questionnaire was administered with computer-assisted personal interviewing (CAPI) through face-to-face interviews at participants' homes.
Groups:
- Overall Sample: Population aged 15 years or more from 12 European countries
Period: Overall Study
Arm/Group | Overall Sample
Started | 11902
Completed | 11902
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Sample
Number analyzed (Participants) | 11902
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 572
  Between 18 and 65 years | 9283
  >=65 years | 2047
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (17.1)
Age, Customized [Median (Full Range); unit: years] | 46 [15 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6270
  Male | 5632
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Bulgaria | 1050
  United Kingdom | 1013
  France | 1018
  Germany | 1031
  Greece | 1000
  Ireland | 941
  Italy | 1059
  Latvia | 1022
  Poland | 724
  Portugal | 1000
  Romania | 1018
  Spain | 1026

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Daily Exposure to Secondhand Smoke (SHS) in Indoor Settings
Description: Exposure to secondhand smoke (SHS) is assessed among non-smokers and indicates the general daily exposure (during a working day and during a non-working day) to SHS in indoor settings (i.e., at home, at workplace, in public and private transports and in other indoor settings). SHS exposure is self-reported and is assessed through a face-to-face interview at baseline (thus representing current exposure at interview).
Time Frame: Baseline
Population: Non-smokers (i.e., never and former smokers) aged 15 years or more from 12 European countries
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Sample
Number analyzed (Participants) | 8562
Participants | 2888

2. Primary Outcome: Prevalence of Exposure to Secondhand Aerosol (SHA) From Electronic Cigarettes
Description: Exposure to secondhand aerosol (SHA) is assessed among electronic cigarette non-users and indicates the general daily exposure (during a working day and during a non-working day) to SHA in indoor settings (i.e., at home, at workplace, in public and private transports and in other indoor settings). SHA exposure is self-reported and is assessed through a face-to-face interview at baseline (thus representing current exposure at interview).
Time Frame: Baseline
Population: Electronic cigarette non-users (i.e., never or former users) aged 15 years or more from 12 European countries
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Sample
Number analyzed (Participants) | 11604
Participants | 1858

3. Secondary Outcome: Prevalence of Never, Current and Former Smokers
Description: Cigarette consumption is assessed at baseline (thus representing current use at interview) through self-reported questions on lifetime use. Never smokers were defined as participants who had never smoked or had smoked less than 100 cigarettes in their lifetime. Smokers were defined as participants who reported smoking at least 100 cigarettes (including hand-rolled cigarettes) during their lifetime. Current smokers were smokers who reported smoking at the time they participated in this survey, while former smokers were smokers who stopped smoking by the time they participated in this survey.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Sample
Number analyzed (Participants) | 11902
Participants
  Never smokers | 6513
  Former smokers | 2049
  Current smokers | 3340

4. Secondary Outcome: Prevalence of Never, Current and Former Electronic Cigarette Users
Description: Electronic cigarette use is assessed at baseline (thus representing current use at interview) through self-reported questions on lifetime use. Current electronic cigarette users were defined as those who reported using the electronic cigarette occasionally (5 days or less) or regularly (more than 5 days) in the last 30 days. Former users of electronic cigarette were those who reported using it in the part but not over the last 30 days.
Time Frame: Baseline
Population: Participants with available information on electronic cigarette use
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Sample
Number analyzed (Participants) | 11876
Participants
  Never users | 11299
  Former users | 305
  Current users | 272

ADVERSE EVENTS:
Arm/Group | Overall Sample
All-Cause Mortality (participants affected / at risk) | 0/11902
Serious Adverse Events (participants affected / at risk) | 0/11902
Other Adverse Events (participants affected / at risk) | 0/11902

LIMITATIONS AND CAVEATS:
* limitations inherent to the cross-sectional study design
* there are some differences of sampling in the study countries
* there was relatively small sample size in each country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT02928536/Prot_SAP_000.pdf